CLINICAL TRIAL: NCT06910774
Title: Analysis of Peripheral Serotonin Levels in a Control Cohort
Acronym: ASPECT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/0033
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: No Condition : to Establish Reference Serum Serotonin Levels in a Control Cohort
Keywords: serotonin (5-HT); tryptophan; control cohort; age; sex; iron status
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The remaining blood samples from the samples taken as part of the treatment will be the subject of a biological collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- control cohort: * Adult patients aged ≥ 18 years
  * Who have undergone a blood draw at CHSF during the recruitment period
  * With hemoglobin, white blood cell, and platelet counts within the laboratory's normal ranges
  * With a C-reactive protein (CRP) level < 30 mg/L
  Interventions: Other: Dosage of serotonin and tryptophan metabolites levels in serum

INTERVENTIONS:
Other: Dosage of serotonin and tryptophan metabolites levels in serum — These measurements will be performed on residual blood samples in the laboratory, after blood collection carried out as part of routine care. Patients will not need to undergo an additional blood draw.

SUMMARY:
The goal of this observational study is to measure serotonin levels in in a control cohort.

The main question aims to determine the mean serum serotonin level in a cohort of adult controls, based on age and sex.

This will allow for the establishment of reference values. We will also measure the different metabolites of tryptophan. These measurements will be performed on residual blood samples in the laboratory, after blood collection carried out as part of routine care. Thus, patients will not need to undergo an additional blood draw.

DETAILED DESCRIPTION:
Serotonin (5-HT or 5-hydroxytryptamine) is a monoamine primarily recognized for its role as a neurotransmitter in the central nervous system (CNS). It is synthesized from tryptophan, which is also essential for the production of metabolites in the kynurenine and indole families.

However, serotonin's functions extend beyond the CNS: various peripheral tissues have the capacity to produce and/or utilize serotonin locally, forming systems referred to as "micro-serotonergic." Among serotonin's peripheral roles, it has been demonstrated to positively influence erythropoiesis and red blood cell survival, iron metabolism, skin pigmentation, as well as placental and embryonic development during pregnancy.

In humans, there is no established standard for blood serotonin levels. It is known that, aside from major events, an individual's serotonin levels remain stable throughout life, but it is likely that blood serotonin levels depend on age and sex.

We aim to establish a cohort of adult control patients, for whom we will measure serum serotonin and the different metabolites of tryptophan, to analyze whether serotonin varies according to sex and age, and to determine its average serum levels.

Preliminary data from the laboratory suggest a role for serotonin in iron metabolism. Therefore, as a secondary objective, we also intend to perform an iron status assessment in control patients to analyze whether there are variations in iron parameters based on serotonin levels.

This cohort could also serve as a comparison point for future studies of serum serotonin levels in pathological conditions or during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged ≥ 18 years
* Who have undergone a blood draw at CHSF during the recruitment period
* With hemoglobin, white blood cell, and platelet counts within the laboratory's normal ranges
* With a C-reactive protein (CRP) level < 30 mg/L

Exclusion Criteria:

* Patients informed about the study who decline participation
* Patients with a current diagnosis or history of psychiatric disorders
* Patients on antidepressants or narcotics at the time of sampling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is a control cohort. We will include adult patients aged 18 years or older who have undergone a blood draw at CHSF during the recruitment period. Eligible participants must have hemoglobin, white blood cell, and platelet counts within the laboratory's normal ranges, and a C-reactive protein (CRP) level below 30 mg/L.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2025-06-23 (Actual); Primary Completion 2025-11-16 (Actual); Study Completion 2025-11-16 (Actual)

PRIMARY OUTCOMES:
Serotonin | at day 0
  Measurement of serotonin levels in serum (HPLC: high performance liquid chromatography)

SECONDARY OUTCOMES:
Tryptophan metabolites | at day 0
  Measurement of tryptophan metabolites levels in serum (HPLC: high performance liquid chromatography)

CONTACTS AND LOCATIONS:
Overall Officials: Guillemette FOUQUET, MD, Principal Investigator — Centre Hospitalier Sud Francilien
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France, France

IPD SHARING:
Plan to Share IPD: No